CLINICAL TRIAL: NCT03331029
Title: Assessment of Left Atrial Mechanical Function With a True 3D Ultrasound Array and Comparison With the Transthoracic and Transesophageal Echocardiography: A Single Center Interventional Study in Patients Scheduled for Ablation Procedure
Brief Title: Assessment of Left Atrial Mechanical Function With a True 3D Ultrasouns Arry and Comparison With the Transthoracic and Transesophageal Echocardiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinik Hirslanden, Zurich (Other)
Responsible Party: Principal Investigator, Werner Baulig, PD Dr. med. Werner Baulig, Senior consultant, Klinik Hirslanden, Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KlinikHirslanden
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Comparison of 3D Monitored Changes of Left Atrial Volume Before and After Ablation With Conventional Transesophageal Echocardiography
Keywords: 3 D Ultrasound, left atrium, Mitral inflow velocity, systolic and diastolic ventricular function
MeSH Terms: conditions — Systolic Murmurs

STUDY DESIGN:
Intervention Model Description: Single Center interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- transesophageal echocardiography (Other): Comparison of 3D Ultrasound with transesophageal echokardiography
  Interventions: Device: transesophageal investigation

INTERVENTIONS:
Device: transesophageal investigation — Comparison of 3D ultrasound with transesophageal echocardiography

SUMMARY:
Chronic atrial fibrillation is a challenging arrhythmia requiring additional radiofrequency ablation besides pulmonary vein isolation. Atrial contractility in these patients is often impaired. Until now mapping catheters were used on virtual geometry maps of left atrium. However, changes in atrial volume cannot be assessed with these systems Assessments of atrial volumes with echocardiography relies on 2D and 3D measurements and modeling. The AcQMapTM 3D High Resolution Imaging and Mapping System (AcQMap) has a unique 3D array of ultrasound crystals, which can measure true 3D dimensions of the heart chamber. For the first time, true atrial volumes can be measured. Changing from atrial fibrillation to sinus rhythm causes changes in atrial volume and might be associated with quantitative systolic and diastolic function of the left ventricle measured with the Transesophageal Echocardiography.

DETAILED DESCRIPTION:
Comparison of true 3D atrial volume changes to TEE and TTE findings as well as atrial pressure curves during left heart catheterization. Changing from atrial fibrillation to sinus rhythm causes changes in atrial volume and might be associated with quantitative systolic and diastolic function of the left ventricle measured with the Transesophageal Echocardiography

Measurement of true left atrial ejection fraction and comparison to 2D echocardiographic parameters such as transesophageal measured flow velocity of the mitral inflow tract, pulmonary vein flow, the left atrial appendage flow

Inclusion:

Patients undergoing electrophysiological study with the AcQmap System Age ≥18 years and signed informed consent German speaking

Exclusion:

Mechanical mitral valve Contraindication for left atrial ablation procedure such as: Intra-cardiac clot, Pregnancy

Data collection of ultrasound dimensions of left atrium, left atrial pressure and TEE is performed simultaneously under the following conditions:

1. Fixed heart rate by atrial pacing
2. Apnea initiated at the end of expiration (apnea endexp)
3. With and without complete atrioventricular bloc Under these conditions pressure volume loops are monitored. Simultaneously mitral annulus velocity (septal and lateral), pulmonary vein flow, left atrial appendage flow (max. A and V velocity) and LAA volume (average of 4 planes) are measured

The AcQMap Catheter consists of 6 splines with 48 electrodes and ultrasound crystals, which form a true 3D array of about 2 cm diameter. The catheter can be collapsed for introduction over a sheet into the right or left atrium and is used to record electrical bio potentials of the atrium. Besides each electrode is an ultrasound crystal, which measures the distance to the atrial wall at a sample rate 100000/min a ultrasound based anatomy of the atrium is constructed. The procedure of introduction the AcQMap catheter is in the right or left atrium is the same as it is performed with the standard devices for mapping and treating the atrial fibrillation in humans.

Analysis of changes in the collected data before and after ablation procedure is performed using unpaired t-test and non-parametric interrogation (Wilcoxon and Mann-Whithey U test) where otherwise appropriate (spss v 16, SPSS Chicago, IL, USA). Normal distributed date will be presented as mean ±SD and 95% confidence interval (CI95) and not normal distributed data will be presented as median and interquartile range (ICR). For repeated measures ANOVA will be used to estimate between-subject's variation and within-subject variation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing electrophysiological study with the AcQmap System
* Age ≥18 years and signed informed consent
* German speaking

Exclusion Criteria:

* Mechanical mitral valve
* Contraindication for left atrial ablation procedure such as: Intra-cardiac clot,
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Mitral flow velocity | 1 hour
changes in pulmonary vein flow | 1 hour
changes in left atrial appendage flow | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Werner Baulig, MD, Principal Investigator — Klinik Im Park, Hirslanden, Zürich, Switzerland
Locations (1):
- Klinik Im Park, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No